CLINICAL TRIAL: NCT01408953
Title: A Therapeutic Trial of Intralesional Bevacizumab in Patients With Non-pedunculated Keloids
Brief Title: Therapeutic Study of Bevacizumab Injection Directly Inside the Keloid Tissue
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Very low accrual rate.
Sponsor: Tirgan, Michael H., M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tirgan 11-03
Record Dates: First submitted 2011-07-29; First posted 2011-08-03 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Keloid
Keywords: Keloid
MeSH Terms: conditions — Keloid | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bevacizumab for all patients (Experimental): This is a single arm trial. All patients receive treatment with bevacizumab.
  Interventions: Biological: bevacizumab

INTERVENTIONS:
Biological: bevacizumab — Bevacizumab will be diluted with 0.9% Sodium Chloride to achieve a concentration of 1 mg/0.3 ml. Bevacizumab will be injected inside ONE keloid tissue to result in a visual expansion of the keloid. Only 1 mg of bevacizumab is injected inside ONE keloid. The injections will be repeated every 14 days. Patients will receive maximum of 12 injections only.
  A log will be kept for each patient indicating the date and the dose of bevacizumab that was delivered to each patient.
  Other Names: Avastin is the brand name for bevacizumab.

SUMMARY:
Keloid is chronic skin conditions that results in formation of tumor like growths on the skin. Despite its benign nature, keloid can cause severe aesthetic and, in some cases, functional problem which negatively impacts person's quality of life.

Keloids do not regress on their own and results of most available treatments such as surgery, injecting keloids with steroids, chemotherapy injections, or even radiation therapy, have mostly proven disappointing.

Some laboratory studies have shown that there is excessive amount of a protein called "vascular endothelial growth factor (VEGF)" in keloid tissue. This may play role in the formation and evolution of keloid.

Bevacizumab is a drug that works by targeting vascular endothelial growth factor (VEGF) which helps new blood vessels form. Without new blood vessels, the growth of the keloid may be slowed

Based on presence of excess amount of VEGF in keloid tissue, we hypothesize that bevacizumab will be effective in treatment of keloids. This exploratory clinical trial is to confirm or reject this hypothesis.

DETAILED DESCRIPTION:
Sixty Eligible patients will be enrolled in the study. This will be a two stage design trial.

In stage I of the trial, 21 patients will be treated with intralesional bevacizumab. Keloids that fail to respond to 4 injections will not be treated any longer with bevacizumab and all such patients will be removed from the trial.

If 5 or more patients show some degree of objective response to treatment in at least one treated keloid, the trial will continue to enroll another 45 patients to a total of 66 patients, otherwise, the trial will stop in its entirety.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical Diagnosis of a flat keloid.
2. Age 18 to 50
3. A signed informed consent document (ICD)
4. Able and willing to receive bevacizumab

Women of child-bearing potential must have a negative pregnancy test during screening. The effects of bevacizumab on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

1. Pedunculated Keloid
2. Diastolic Blood pressure of 90 mm Hg or above
3. History of any degree of Hypertension, even medically controlled hypertension
4. History of any form of cardiovascular disease or stroke
5. History of any form of thromboembolic event
6. History of renal dysfunction or proteinuria
7. History of recent (past 12 month) or planned (next 3 months) major surgery,
8. Men and women who plan to have children within 6 months of their last treatment
9. Psychological Illness that may result in non compliance with treatment
10. Pregnancy and Breast Feeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this trial is to demonstrate the response rate of non-pedunculated keloids to bevacizumab. | 1 year
  The primary objective of this trial is to demonstrate the efficacy of bevacizumab in patients with non-pedunculated keloids. Patients will be followed for one year since their last bevacizumab to assess post-therapy duration of response as well as the rate of recurrence.

SECONDARY OUTCOMES:
The secondary endpoint of this trial is to demonstrate the rate of AE and SAE following intralesional Injections of bevacizumab. | 1 Year
  The secondary objective of this trial is to demonstrate safety of intralesional bevacizumab. Patients will be followed for one year after their last bevacizumab to assess safety of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Tirgan, MD, Study Chair — Keloid Research Foundation
Locations (1):
- Michael H. Tirgan, MD, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Only two patients were treated on this study, neither responded. The study was closed due to difficulties in accruing patients.